CLINICAL TRIAL: NCT02397083
Title: Phase II Study of the Levonorgestrel Intrauterine Device Alone or in Combination With the mTORC1 Inhibitor, Everolimus, for the Treatment of Complex Atypical Hyperplasia and Stage Ia Grade 1 Endometrial Cancer
Brief Title: Levonorgestrel-Releasing Intrauterine System With or Without Everolimus in Treating Patients With Atypical Hyperplasia or Stage IA Grade 1 Endometrial Cancer
Acronym: LEVER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0944; NCI-2015-00919 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0944 (Other: M D Anderson Cancer Center); P50CA098258 (NIH)
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Atypical Endometrial Hyperplasia; FIGO Grade 1 Endometrial Endometrioid Adenocarcinoma; FIGO Grade 2 Endometrial Endometrioid Adenocarcinoma
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (LIUD) (Experimental): Patients continue treatment with the LIUD for up to 9 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Device: Levonorgestrel-Releasing Intrauterine System
- Arm II (LIUD, everolimus) (Experimental): Patients continue treatment with the LIUD and receive everolimus PO QD on days 1-28. Treatment repeats every 28 days for up to 9 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Other: Laboratory Biomarker Analysis; Device: Levonorgestrel-Releasing Intrauterine System

INTERVENTIONS:
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
  Arms: Arm II (LIUD, everolimus)
Other: Laboratory Biomarker Analysis — Correlative studies
Device: Levonorgestrel-Releasing Intrauterine System — Placed in the uterus
  Other Names: Mirena

SUMMARY:
This randomized phase II trial studies how well levonorgestrel-releasing intrauterine system works when given alone or with everolimus in treating patients with atypical hyperplasia (a pre-cancerous growth of the lining of the uterus) or stage IA grade 1 endometrial cancer. The levonorgestrel-releasing intrauterine system is designed to prevent pregnancy by releasing a hormone called levonorgestrel, which is a type of progesterone. Progesterone is a common type of hormone that is used to prevent pregnancy and may prevent or slow tumor cell growth. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether the levonorgestrel-releasing intrauterine system works better with or without everolimus in treating patients with atypical hyperplasia or stage IA grade 1 endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the efficacy of the levonorgestrel intrauterine device (LIUD) (levonorgestrel-releasing intrauterine system) alone to treat complex atypical hyperplasia or stage Ia grade 1 endometrioid endometrial carcinoma with response rate.

II. Estimate the efficacy of the LIUD in combination with everolimus to treat LIUD-refractory complex atypical hyperplasia or stage Ia grade 1 endometrioid endometrial carcinoma with response rate.

SECONDARY OBJECTIVES:

I. Document the toxicity profile of the levonorgestrel intrauterine device alone or in combination with everolimus using the National Institutes of Health-National Cancer Institute (NIH-NCI) Common Terminology Criteria for Adverse Events version (v) 4.0.

II. Estimate overall survival (OS) and event-free survival (EFS) of patients with complex atypical hyperplasia or stage Ia grade 1 endometrioid endometrial cancer treated with the levonorgestrel IUD alone or in combination with everolimus.

III. Estimate the response duration associated with the levonorgestrel IUD alone or in combination with everolimus in patients with complex atypical hyperplasia or stage Ia grade 1 endometrioid endometrial cancer.

EXPLORATORY OBJECTIVE:

I. Determine if response to therapy can be predicted based on the molecular profile of the tumor, including estrogen-induced genes and relevant pathway members, or by change in gene expression after therapy.

OUTLINE:

First Stage

* If D&C confirms EEC grade 1 or CAH-patient enrolled
* If the patient is found to have stable disease at 3 months continue on to the second stage of the study to be randomized.
* If the patient has a complete response at 3 months; EMB 3 months later to confirm complete response.
* Once complete response confirmed, patient Continues EMB every 6-12 months until disease progression per provider.
* If the patient has progressive disease at 3 months- OFF STUDY Second Stage
* Patients with stable disease at and 3 month EMB, recurrent disease at a subsequent EMB, or entering protocol with outside IUD in place showing stable disease demonstrating progesterone resistance

LIUD Only Arm

* Visits every 3 months
* EMB at 6 months
* if regression/SD: continue on study
* EMB at 9 months and 1 year:
* Off study for PD or D&C at MD's discretion
* SD at 1 year: off study
* CR at 1 year: SOC EMB 3 months later then Q6 months if confirmed CR
* If continuing on study: Q6mo EMB until progression, D&C, or pt./provider decision

LIUD+Everolimus Arm

* If progression at cycle 3, 6, 9:
* Discontinue everolimus, patient taken off study
* CR at cycle 9:
* EMB to confirm response at cycle 12
* If response confirmed -EMB every 6 cycles (6 months)
* Continue evaluations on each cycle day 1
* SD at cycle 9:
* Discontinue everolimus, come off study

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of complex atypical hyperplasia OR, grade 1 endometrioid OR focal grade 2 adenocarcinoma in predominately grade 1 disease endometrial carcinoma on endometrial biopsy or dilation and curettage (D & C) within three months of study enrollment
* Patients with complex atypical hyperplasia OR grade 1 endometrioid adenocarcinoma with stable/persistent disease with LIUD already in place. LIUD must have been in place for at least 3 months
* Prior progesterone treatment is ALLOWED, but a 28 day washout period is required before LIUD placement. If archival tissue is available from prior to any progesterone treatment, the washout period is not needed
* Ability to comply with endometrial biopsies every 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hb) > 9 g/dL
* Total serum bilirubin =< 2.0 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN)
* International normalized ratio (INR) =< 2; factor 10A drawn if patient on anticoagulant Eliquis
* Serum creatinine =< 1.5 x ULN
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L AND fasting triglycerides =< 2.5 x ULN; NOTE: in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Signed informed consent obtained prior to any screening procedures

Exclusion Criteria:

* Patients with grade 2-3 endometrioid, uterine serous, clear cell, mucinous, squamous, transitional cell, sarcomas, or carcinosarcoma histology
* Evidence of extrauterine spread of disease on imaging or during surgical evaluation
* Patients who have prior therapy with everolimus or any other mammalian target of rapamycin (mTOR) inhibitor
* Patients currently receiving anticancer therapies (including chemotherapy, radiation therapy, hormonal, or antibody-based therapy); prior treatment should have a washout period of 28 days or 4 1/2 half-lives (7 days), whichever is shorter
* Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus)
* Known intolerance or hypersensitivity to progesterone or its excipients
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus (e.g., inability to take oral medication or a requirement for intravenous [IV] alimentation, prior surgical procedures affecting absorption, malabsorption syndrome, and active peptic ulcer disease) are excluded; subjects with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction are also excluded, as are any patients who cannot swallow the capsule whole
* Uncontrolled diabetes mellitus as defined by glycosylated hemoglobin (HbA1c) > 8% despite adequate therapy; patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary
* Patients who have any severe and/or uncontrolled medical conditions such as: a) unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction =< 6 months prior to start of everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease; b) symptomatic congestive heart failure of New York Heart Association class III or IV; c) active (acute or chronic) or uncontrolled severe infection (not responding to antibiotics), liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis (i.e. quantifiable hepatitis B virus-deoxyribonucleic acid [HBV-DNA] and/or positive hepatitis B surface antigen [HbsAg], quantifiable hepatitis C virus-ribonucleic acid [HCV-RNA]); d) known severely impaired lung function (spirometry and diffusing capacity of the lung for carbon monoxide [DLCO] 50% or less of normal and oxygen [O2] saturation 88% or less at rest on room air); e) active, bleeding diathesis
* Chronic treatment with corticosteroids or other immunosuppressive agents; topical or inhaled corticosteroids are allowed
* Patients who have a known history of human immunodeficiency virus (HIV) seropositivity
* Patients who have received live attenuated vaccines within 1 week of start of everolimus and during the study; patient should also avoid close contact with others who have received live attenuated vaccines; examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guerin (BCG), yellow fever, varicella and TY21a typhoid vaccines
* Other malignancies within the past 3 years except for basal or squamous cell carcinoma of the skin
* Active (acute or chronic) or uncontrolled severe infections (not responding to antibiotics), including acute pelvic inflammatory disease
* Congenital or acquired uterine anomaly which distorts the uterine cavity
* Genital actinomycosis
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Women who are pregnant or nursing (lactating) women
* Women of child-bearing potential (WOCBP), defined as women physiologically capable of becoming pregnant, must use one additional highly effective methods of contraception in addition to the LIUD during the study and 8 weeks after; acceptable effective contraception methods include combo of the following: a) barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository; b) total abstinence or; c) male/female sterilization; women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation > six weeks prior to randomization; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential
* Women who are on contraindicated medications to everolimus must have confirmation from their physician that they may change or discontinue the medication if randomized to the LIUD + everolimus arm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Response rate (levonorgestrel intrauterine device [LIUD] alone) | At 3 months
  Estimated with a 2-sided 90% confidence interval.
Response rate (levonorgestrel intrauterine device [LIUD] alone) | 6 months
  Estimated with a 2-sided 90% confidence interval.
Response rate for levonorgestrel intrauterine device (LIUD) alone or in combination with everolimus after LIUD failure (i.e., failure to achieve complete response after initial 3 months of LIUD alone) | 6 months
  Fisher's exact test will be used to compare response rates by 6 months between the LIUD alone arm and the LIUD plus everolimus arm. Estimated on each arm with a 2-sided 90% confidence interval.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 11 years
  Tabulated by treatment arm, severity, and relationship to study drug.
Progression free survival | Up to 11 years
  Estimated using the Kaplan-Meier product-limit estimator. The log-rank test will be used to compare treatment arms.
Overall survival | Up to 11 years
  Estimated using the Kaplan-Meier product-limit estimator. The log-rank test will be used to compare treatment arms.
Response duration | Up to 4 weeks after completion of study treatment
  Estimated using the Kaplan-Meier product-limit estimator. The log-rank test will be used to compare treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (18):
- United States (18):
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Queen's Medical Center, Honolulu, Hawaii
  - Covenant HealthCare Mackinaw, Saginaw, Michigan
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Northwell Health, New Hyde Park, New York
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - MD Anderson in The Woodlands, Conroe, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org